CLINICAL TRIAL: NCT03795766
Title: Prevalence and Predictors of Nausea and Vomiting After Gynecologic Surgery: a Cross-section Study
Brief Title: Nausea and Vomiting After Gynecologic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Other Study IDs: GY-PONV
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Nausea and Vomiting; Gynecologic Surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgeries for gynecologic disease — All patients accept surgeries for gynecologic disease.

SUMMARY:
In this cross-section study, all patients in the gynecologic ward of Peking Union Medical College Hospital will accepted a survey about the prevalence and severity of nausea and vomiting according to visual analogue scale and WHO classification. Epidemiological, surgical, anaesthetic characteristics and post-operative treatment are considered as predictors for the post-operative nausea and vomiting. The primary objective is the incidence of nausea and vomiting. The secondary objective is the possible predictors of nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Elective surgeries for gynecologic disease
* Good performance status
* Signed an approved informed consents
* Post-operative stay 72 hours or longer

Exclusion Criteria:

* Emergency surgeries
* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients accept elective surgeries for gynecologic disease with good performance status.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-operative nausea and vomiting | 72 hours post-operative
  Incidence of post-operative nausea and vomiting

SECONDARY OUTCOMES:
Severity of post-operative nausea and vomiting by visual analogue scale | 72 hours post-operative
  Severity of post-operative nausea and vomiting according to the visual analogue scale. In th scale, 0 denotes none, 10 denotes the most severe conditions. The scale will be judged by the patients.
Severity of post-operative nausea and vomiting by World Health Organization classification | 72 hours post-operative
  Severity of post-operative nausea and vomiting according to World Health Organization (WHO) classification. In WHO classfication, I denotes none, II, III and IV denote mild, moderate and severe conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided